CLINICAL TRIAL: NCT06258811
Title: Neoadjuvant Immunochemotherapy With Tislelizumab, Albumin Paclitaxel and Cisplatin Followed by Standard Therapy Versus Standard Therapy for Locally Advanced Oral Squamous Cell Carcinoma, a Multicenter Randomized Phase 3 Trial
Brief Title: Neoadjuvant Immunochemotherapy for LAOSCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lai-ping Zhong (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other); Central South University (Other); Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, Lai-ping Zhong, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TopHill
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Oral Squamous Cell Carcinoma; Locally Advanced Head and Neck Carcinoma
Keywords: Oral squamous cell carcinoma; Neoadjuvant immunochemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to experimental or control arm. Experiment arm: neoadjuvant immunochemotherapy (2 cycles, and 21 days each cycle, 260mg/m2 albuminpaclitaxel intravenously on day 1 and day 22, with 75mg/m2 of cisplatin and 200mg of tislelizumab) + radical surgery + adjuvant therapy (radiation/chemoradiation followed by 200mg of tislelizumab, every 3 weeks for one year) Control arm: standard therapy of radical surgery +adjuvant therapy (radiation/chemoradiation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Neoadjuvant immunochemotherapy (albumin paclitaxel+cisplatin+tislelizumab) + radical surgery + adjuvant therapy (radiation/chemoradiation + tislelizumab maitainance)
  Interventions: Drug: albumin paclitaxel, cispatin, tislelizumab
- Control arm (No Intervention): Standard therapy of radical surgery +adjuvant therapy (radiation/chemoradiation)

INTERVENTIONS:
Drug: albumin paclitaxel, cispatin, tislelizumab — Neoadjuvant immunochemotherapy (2 cycles, and 21 days each cycle, 260mg/m2 albumin paclitaxel intravenously on day 1 and day 22, with 75mg/m2 of cisplatin and 200mg of tislelizumab) + radical surgery + adjuvant therapy (radiation/chemoradiation followed by 200mg of tislelizumab, every 3 weeks for one year)
  Arms: Experimental arm

SUMMARY:
To evaluate the prognostic efficacy of neoadjuvant immunochemotherapy with tislelizumab, albumin paclitaxel and cisplatin followed by radical surgery and adjuvant therapy compared with standard therapy for patients with locally advanced and resectable oral squamous cell carcinoma.

DETAILED DESCRIPTION:
Neoadjuvant therapy (NAT) is regarded as an effective way to reduce or downgrade the locally advanced or aggressive cancers, and to improve the chance of eradication of the locoregional lesions by radical surgery and/or radiotherapy. However, there are still debates on the clinical value of NAT for patients with locally advanced oral squamous cell carcinoma (LAOSCC). In a series of clinical trials on neoadjuvant therapy for LAOSCC have been carried out by our research group, the pathological efficacy of neoadjuvant immunochemotherapy is superior to neoadjuvant immunotarget therapy, neoadjuvant chemotarget therapy, or neoadjuvant chemotherapy. And in the neoadjuvant immunochemotherapy clinical trial (NCT04473716), the results of the safety and efficacy of neoadjuvant regimen showed that the neoadjuvant regimen of immunochemotherapy was well tolerated, with an MPR rate of 60% and 2-year OS of 90%, which were better than previously reported patients receiving standard treatment for LAOSCC. However, limited to single-arm clinical trial, the patients with LAOSCC benefit from neoadjuvant immunochemotherapy for survival, randomized controlled trials with larger sample size are needed. The aim of present trial is to evaluate the prognostic efficacy of 2-year survival rate in patients with LAOSCC receiving neoadjuvant immunochemotherapy with tiralizumab, albumin paclitaxel and cisplatin followed by radical surgery and adjuvant therapy compared with standard therapy.

The patients with LAOSCC would receive NAT with tiralizumab, albumin paclitaxel and cisplatin followed by radical surgery and adjuvant therapy (the experimental group) or radical surgery and adjuvant therapy (the control group). A total number of 134 patients will be recruited. Neoadjuvant immunochemotherapy: for the patients who are randomly assigned to the experimental group, the palpable edges of the primary lesion (both the longest and shortest axis) would be marked before NAT by at least four points, which is 0.5cm away; 260mg/m2 albuminpaclitaxel intravenously on day 1 and day 22, with 75mg/m2 of cisplatin at an hour interval and 200mg of tislelizumab at an hour interval will be performed. NAT will be given every 3 weeks for 2 cycles, unless there is disease progression, unacceptable toxic effects, or withdrawal of consent by the patients. Surgery will be performed within 2 weeks after completion of NAT. Surgery: Radical resection of the primary lesion and full neck dissection with proper reconstruction will be performed. The safety margins of the primary lesion are 1.0-1.5cm far away from the palpable margins of the lesion; for patients who received NAT, the safety margins are 1.0cm away from the marks that were placed before NAT, to ensure the same extent surgery in both groups. Post-operative adjuvant therapy: radiotherapy will be arranged 4 to 6 weeks after surgery. Routine external beam radiotherapy, will be performed, and the dose is 1.8-2Gy/day, 5 days/week for 6 weeks, and totally 54-60Gy, in the patient with high risk features, concurrent chemotherapy with cisplatin of 80mg/m2 will be used; in the experimental group, adjuvant maintaining therapy of 200mg of tislelizumab, every 3 weeks, for one year will be used. A complete medical history will be obtained and tumor assessment will be performed at baseline. Clinical tumor response will be assessed by clinical evaluation, imaging evaluation will be characterized according to the criteria of response evaluation criteria in solid tumors (version 1.1) before surgery. Post-operative pathological response will be assessed by post-operative pathological examination. Patients will be followed-up by every three months in the first 2 years, every six months in the next 3-5 years, and once a year thereafter until death or data censoring. Overall survival will be calculated from the date of randomization to the date of death; event free survival will be calculated from the date of randomization to local recurrence, regional recurrence, distant metastasis, disease progress, or death; disease free survival will be calculated from the date of randomization to tumor recurrence or distant metastasis or death from any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-1
2. Histopathological diagnosis of oral squamous cell carcinoma (including tongue, gums, cheek, floor of mouth, hard palate, and posterior molar region)
3. Primary tumor with a clinical stage of III/IVA (T1-2/N1-2/M0 or T3-4a/cN0-2/M0, AJCC 2018)
4. Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
5. Blood routine: white blood cells (WBCs) >3,000/mm3, hemoglobin >8 g/L, platelets >80,000/mm3
6. Liver function: alanine amino transferase/aspartate amino transferase (ALAT/ASAT) <2.5 times the upper limit of normal and bilirubin <1.5 times the upper limit of normal
7. Renal function: Serum creatinine <1.5 times the upper limit of normal
8. Coagulation function: INR、PT、APTT<1.5 times the upper limit of normal
9. Signed the informed consent form

Exclusion Criteria:

1. Unresolved grade 2 [(Common Terminology Criteria for Adverse Events (CTCAE 5.0)] or higher toxic reactions caused by previous anticancer treatments
2. Known allergic reaction (grade 3-4) to any ingredients or excipients of the therapy
3. Known history of malignancy, unless been cured and no recurrence for 5 years
4. Known history of radiation to head and neck
5. Active severe clinical infection (> National Cancer Institute (NCI)-CTCAE version 5.0 grade 2 infection)
6. Obvious cardiovascular abnormalities [such as myocardial infarction, superior vena cava syndrome, grade 2 or higher heart disease diagnosed according to the New York Heart Association (NYHA) classification 3 months before enrollment]
7. Patients receiving immunology-based treatment for any reason
8. Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy
9. Pregnant or lactating women
10. Known active hepatitis B or C. Active hepatitis B is defined as a known HBsA positive with HBV DNA≥500 IU/mL. Active hepatitis C is defined as a known hepatitis C antibody positive and a known amount of hepatitis C virus HCV RNA results greater than the lower limit of detection. The presence of other serious liver diseases, including chronic autoimmune liver disease, primary biliary cirrhosis or sclerosing cholangitis, alcoholic liver disease, or non-alcoholic steatohepatitis (NASH)
11. Complicated with severe, uncontrolled infection or known human immunodeficiency virus (HIV) infection, or diagnosed as acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or history of allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or solid organ transplantation
12. Participation in other clinical trials within 30 days before enrollment
13. Other situations that the investigator considers unsuitable with respect to participating in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of 2-year event-free survival | 2 years
  Event free survival is calculated from the date of randomization to local recurrence, regional recurrence, distant metastasis, disease progress, or death. The rate of 2-year event free survival is reported as the percentage of patients who are event free survival for 2 years from the date of randomization.
Rate of 2-year overall survival | 2 years
  Overall survival is calculated from the date of randomization to death. The rate of 2-year overall survival is reported as the percentage of patients who are overall survival for 2 years from the date of randomization.

SECONDARY OUTCOMES:
Rate of 2-year disease-free survival | 2 years
  Disease free survival is calculated from the date of randomization to local recurrence, locoregional recurrence, distant metastasis, or death. The rate of 2-year disease free survival is reported as the percentage of patients who are disease free survival for 2 years from the date of randomization.
Rate of major pathological response | 6 months
  Major pathological response is based on the pathological examination on the post-operative specimens after neoadjuvant immunochemotherapy. The rate of major pathological response is reported as the percentage of patients who have major pathological response after NAT.

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, MD, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after completion of the trial, for 6 months.
Access Criteria: Access to IPD data can be obtained upon scientifically sound request from the study PI, who will contact the Clinical Research Unit, Huashan Hospital, Fudan University. Access will be released after the approval from the Clinical Research Unit.